CLINICAL TRIAL: NCT02285062
Title: Phase 3 Randomized, Double-Blind, Placebo Controlled, Multicenter Study to Compare the Efficacy and Safety of Lenalidomide (CC-5013) Plus R-CHOP Chemotherapy (R2-CHOP) Versus Placebo Plus R-CHOP Chemotherapy in Subjects With Previously Untreated Activated B-cell Type Diffuse Large B-cell Lymphoma
Brief Title: Efficacy and Safety Study of Lenalidomide Plus R-CHOP Chemotherapy Versus Placebo Plus R-CHOP Chemotherapy in Untreated ABC Type Diffuse Large B-cell Lymphoma
Acronym: ROBUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-DLC-002; 2013-004054-21 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: R-CHOP chemotherapy; DLBCL front line therapy; gene expression profiling (GEP) activated B-cell (ABC) type DLBCL biomarkers; Activated B-Cell (ABC) type; Diffuse Large B-Cell Lymphoma, not otherwise specified; Diffuse Large B-Cell Lymphoma, associated with chronic inflammation; Diffuse Large B-Cell Lymphoma, Epstein-Barr virus positive (EBS+) of the elderly; Diffuse Large B-Cell Lymphoma, T-cell / histiocyte-rich
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Limb-girdle muscular dystrophy, type 2C | interventions — Lenalidomide; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R2-CHOP (Experimental): Lenalidomide plus R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone)
  Interventions: Drug: lenalidomide; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: prednisone; Drug: vincristine
- R-CHOP (Active Comparator): Placebo plus R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone)
  Interventions: Drug: Placebo; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: prednisone; Drug: vincristine

INTERVENTIONS:
Drug: lenalidomide
  Arms: R2-CHOP
Drug: Placebo
  Arms: R-CHOP
Drug: Rituximab
Drug: Cyclophosphamide
Drug: Doxorubicin
Drug: prednisone
Drug: vincristine

SUMMARY:
To evaluate the efficacy and safety of lenalidomide, rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R2-CHOP) chemotherapy versus placebo, rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (placebo-R-CHOP) chemotherapy in patients who have previously untreated ABC type DLBCL.

DETAILED DESCRIPTION:
This research study is for patients with newly diagnosed Diffuse Large B-cell Lymphoma (DLBCL) of the activated B-cell (ABC) type who have not yet been treated. DLBCL is a cancer of a type of blood cell called B-lymphocytes. B lymphocytes are part of the body's immune system. There are different types of DLBCL. About a third of newly diagnosed DLBCL cancers are the ABC type. It has been observed that treatment does not work as well for patients with the ABC type compared to patients with other DLBCL types who receive standard treatment. However, at this time both ABC type and other DLBCL type patients receive the same standard treatments.

Patients with DLBCL who are otherwise healthy are usually treated first with the chemotherapy drug combination called R-CHOP. The drugs in this combination are "R" for rituximab, "C" for cyclophosphamide, "H" for doxorubicin which has a chemical name of hydroxydaunomycin, "O" for vincristine which has a trade name of oncovin, and "P" for prednisone. Depending on the local practice where you are treated, R-CHOP may be given for 6 or 8 cycles. A cycle could lasts for 14 or 21 days. The R-CHOP drug combination is approved for the treatment of DLBCL of all types, including ABC type. R-CHOP is standard care.

This study will test the standard R-CHOP21 against R-CHOP21 plus lenalidomide. The purpose is to see whether adding lenalidomide works better and is as safe as R-CHOP by itself. This study is only for patients with ABC type DLBCL who have not yet been treated. Lenalidomide is not approved for use in DLBCL. Its use in this disease is experimental. In this study, the experimental treatment is lenalidomide + R-CHOP21 x 6.

This study will use a gene expression profile (GEP) test to see if a patient has the ABC type. The results of this GEP test affect whether you may be treated on this study. Because the performance of this test has not been proven, it is for investigational use only, and is still under development. This means the GEP test is an experimental test.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven Diffuse Large B-Cell Lymphoma of the Activated B-Cell type
2. Newly diagnosed, previously untreated Diffuse Large B-Cell Lymphoma
3. Measurable Diffuse Large B-Cell Lymphoma disease by Computed Tomography (CT) / Magnetic Resonance Imagining (MRI) scans
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
5. Age 18 - 80 years; age > 80 allowed at investigator discretion if performance status ≤ 1; and each organ system score ≤ 2 using cumulative illness rating scale (CIRS)

Exclusion Criteria:

1. Diagnosis of lymphoma histologies other than Diffuse Large B-Cell Lymphoma
2. History of malignancies, other than Diffuse Large B-Cell Lymphoma, unless the patient has been disease free for 5 years or more
3. Known seropositive for, or history of, active Human Immunodeficiency Virus (HIV) Hepatitis B Virus (HBV), Hepatitis C Virus (HCV)
4. Contraindication to any drug in the chemotherapy regimen, and specifically: LVEF (Left Ventricular Ejection Fraction) < 45% or peripheral neuropathy grade 2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (158):
- United States (22):
  - Local Institution - 177, Fayetteville, Arkansas
  - Local Institution - 136, Orange, California
  - Local Institution - 127, Sacramento, California
  - Local Institution - 169, New Haven, Connecticut
  - Local Institution - 128, Hollywood, Florida
  - McFarland Clinic, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Local Institution - 143, Fairway, Kansas
  - Local Institution - 158, Shreveport, Louisiana
  - Center For Cancer And Blood Disorders, Bethesda, Maryland
  - Local Institution - 101, Minneapolis, Minnesota
  - Local Institution - 138, Minneapolis, Minnesota
  - Local Institution - 112, Rochester, Minnesota
  - Local Institution - 103, Durham, North Carolina
  - Local Institution - 161, Philadelphia, Pennsylvania
  - Local Institution - 951, Dallas, Texas
  - Local Institution - 151, Dallas, Texas
  - Local Institution - 146, Salt Lake City, Utah
  - Local Institution - 905, Edmonds, Washington
  - Local Institution - 903, Issaquah, Washington
  - Local Institution - 162, Seattle, Washington
  - Local Institution - 904, Seattle, Washington
- Australia (4):
  - Local Institution - 004, Albury, New South Wales
  - Local Institution - 008, Clayton, Victoria
  - Local Institution - 002, Geelong, Victoria
  - Local Institution - 003, Frankston
- Belgium (4):
  - Local Institution - 301, Brussels
  - Local Institution - 307, Liège
  - Local Institution - 305, Roeselare
  - Local Institution - 303, Sint-Niklaas
- Canada (5):
  - Local Institution - 368, Calgary, Alberta
  - Local Institution - 373, Surrey, British Columbia
  - Local Institution - 366, Saint John, New Brunswick
  - Local Institution - 362, Greenfield Park, Quebec
  - Local Institution - 365, Montreal, Quebec
- China (17):
  - Local Institution - 209, Beijing
  - Local Institution - 206, Beijing
  - Local Institution - 215, Beijing
  - Local Institution - 200, Beijing
  - Local Institution - 211, Changchun
  - Local Institution - 210, Chengdu
  - Local Institution - 213, Chongqing
  - Local Institution - 202, Fuzhou
  - Local Institution - 217, Guangzhou, Guangdong
  - Local Institution - 204, Hangzhou
  - Local Institution - 207, Harbin, Heilongjiang
  - Local Institution - 212, Nanjing
  - Local Institution - 205, Nanjing, Jiangsu
  - Local Institution - 214, Shanghai
  - Local Institution - 219, Suzhu
  - Local Institution - 221, Tianjin
  - Local Institution - 203, Wuhan
- Czechia (5):
  - Local Institution - 376, Brno
  - Local Institution - 377, Hradec Králové
  - Local Institution - 379, Olomouc
  - Local Institution - 380, Prague
  - Local Institution - 378, Prague
- France (7):
  - Local Institution - 576, Bayonne
  - Local Institution - 585, Bordeaux
  - Local Institution - 583, Montpellier
  - Local Institution - 582, Paris
  - Local Institution - 588, Pessac
  - Local Institution - 587, Toulose
  - Local Institution - 581, Vandœuvre-lès-Nancy
- Ireland (2):
  - Local Institution - 893, Dublin
  - Local Institution - 894, Galway
- Israel (7):
  - Local Institution - 273, Beersheba
  - Local Institution - 274, Haifa
  - Local Institution - 272, Jerusalem
  - Local Institution - 275, Kfar Saba
  - Local Institution - 277, Petah Tikva
  - Local Institution - 278, Tel Aviv
  - Local Institution - 270, Ẕerifin
- Italy (29):
  - Local Institution - 690, Terni, Umbria
  - Local Institution - 659, Allessandria
  - Local Institution - 658, Brescia
  - Local Institution - 674, Cuneo
  - Local Institution - 664, Florence
  - Local Institution - 652, Genova
  - Local Institution - 667, Ivrea
  - Local Institution - 684, Meldola
  - Local Institution - 666, Milan
  - Local Institution - 653, Milan
  - Local Institution - 676, Milan
  - Local Institution - 657, Napoli, Campania
  - Local Institution - 655, Novara
  - Local Institution - 685, Padua
  - Local Institution - 686, Pagani
  - Local Institution - 651, Pavia
  - Local Institution - 679, Ravenna
  - Local Institution - 668, Reggio Emilia
  - Local Institution - 683, Rimini
  - Local Institution - 689, Roma
  - Local Institution - 694, Roma
  - Local Institution - 673, Roma
  - Local Institution - 656, Rome
  - Local Institution - 671, Torino
  - Local Institution - 662, Torino
  - Local Institution - 681, Tricase
  - Local Institution - 692, Udine
  - Local Institution - 682, Verona
  - Local Institution - 672, Vicenza
- Japan (12):
  - Local Institution - 508, Chuo-ku, Tokyo
  - Local Institution - 509, Koto-ku, Tokyo
  - Local Institution - 502, Minato-ku, Tokyo
  - Local Institution - 513, Akita
  - Local Institution - 511, Fukuoka
  - Local Institution - 505, Isehara City, Kanagawa
  - Local Institution - 501, Kashiwa
  - Local Institution - 510, Kyoto
  - Local Institution - 506, Minami-Ku, Fukuoka
  - Local Institution - 507, Nagoya
  - Local Institution - 515, Sendai
  - Local Institution - 504, Yamagata
- Netherlands (6):
  - Local Institution - 353, 's-Hertogenbosch
  - Local Institution - 358, Amsterdam
  - Local Institution - 359, Breda
  - Local Institution - 357, Hoofddorp
  - Local Institution - 354, Leeuwarden
  - Local Institution - 350, Schiedam
- New Zealand (2):
  - Local Institution - 240, Christchurch
  - Local Institution - 243, Palmerston
- Portugal (4):
  - Local Institution - 730, Figueira da Foz Municipality
  - Local Institution - 732, Lisbon
  - Local Institution - 729, Lisbon
  - Local Institution - 727, Pragal
- Local Institution - 115, San Juan, Puerto Rico
- Russia (3):
  - Local Institution - 050, Kazan'
  - Local Institution - 052, Moscow
  - Local Institution - 051, Saint Petersburg
- South Korea (4):
  - Local Institution - 830, Gyeonggi-do
  - Local Institution - 826, Seoul
  - Local Institution - 829, Seoul
  - Local Institution - 828, Seoul
- Spain (12):
  - Local Institution - 776, Barcelona
  - Local Institution - 780, Barcelona
  - Local Institution - 796, Cáceres
  - Local Institution - 783, Madrid
  - Local Institution - 785, Madrid
  - Local Institution - 787, Madrid
  - Local Institution - 788, Madrid
  - Local Institution - 797, Salamanca
  - Local Institution - 790, Seville
  - Local Institution - 800, Seville
  - Local Institution - 793, Valencia
  - Local Institution - 802, Valencia
- Switzerland (3):
  - Local Institution - 323, Bellinzona
  - Local Institution - 320, Geneva
  - Local Institution - 321, Winterthur
- Taiwan (3):
  - Local Institution - 253, Niao-Sung Hsiang Kaohsiung County
  - Local Institution - 255, Taichung
  - Local Institution - 252, Taipei, Zhongzheng Dist.
- Turkey (Türkiye) (6):
  - Local Institution - 429, Adana
  - Local Institution - 431, Ankara
  - Local Institution - 430, Antalya
  - Local Institution - 435, Denizli
  - Local Institution - 428, Edirne
  - Local Institution - 432, Istanbul

REFERENCES:
- [Background] Nowakowski GS, Chiappella A, Witzig TE, Spina M, Gascoyne RD, Zhang L, Flament J, Repici J, Vitolo U. ROBUST: Lenalidomide-R-CHOP versus placebo-R-CHOP in previously untreated ABC-type diffuse large B-cell lymphoma. Future Oncol. 2016 Jul;12(13):1553-63. doi: 10.2217/fon-2016-0130. Epub 2016 Apr 18. PMID 27089170
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Nowakowski GS, Chiappella A, Gascoyne RD, Scott DW, Zhang Q, Jurczak W, Ozcan M, Hong X, Zhu J, Jin J, Belada D, Bergua JM, Piazza F, Mocikova H, Molinari AL, Yoon DH, Cavallo F, Tani M, Yamamoto K, Izutsu K, Kato K, Czuczman M, Hersey S, Kilcoyne A, Russo J, Hudak K, Zhang J, Wade S, Witzig TE, Vitolo U. ROBUST: A Phase III Study of Lenalidomide Plus R-CHOP Versus Placebo Plus R-CHOP in Previously Untreated Patients With ABC-Type Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2021 Apr 20;39(12):1317-1328. doi: 10.1200/JCO.20.01366. Epub 2021 Feb 23. PMID 33621109
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent to Treat (ITT) population - all randomized participants. Safety population - all participants that received at least 1 dose of study medication.
Groups:
- Lenalidomide Plus R-CHOP (R2-CHOP): Participants received lenalidomide 15 mg capsules on days 1 to 14 of each 21 day treatment cycle followed by R-CHOP: rituximab 375 mg/m^2 by intravenous (IV) administration on Day 1, doxorubicin 50 mg/m^2 IV on Day 1, vincristine 1.4 mg/m^2 IV on Day 1 (maximum dose of 2.0 mg total), cyclophosphamide 750 mg/m^2 IV on Day 1 and oral or IV prednisone/prednisolone 100 mg on Day 1 to Day 5 of each 21 day treatment cycle for 6 cycles. Treatment continued until completed, unless unacceptable toxicity, treatment change, disease progression, or withdrawal of consent, whichever occurred first. An additional two doses (1 dose per 21-day cycle) of single agent rituximab after the 6 cycles of treatment were completed if considered standard of care per local practice.
- Placebo Plus R-CHOP: Participants received identically matching placebo capsules on days 1 to 14 of each 21 day treatment cycle followed by R-CHOP: rituximab 375 mg/m^2 by intravenous (IV) administration on Day 1, doxorubicin 50 mg/m^2 IV on Day 1, vincristine 1.4 mg/m^2 IV on Day 1 (maximum dose of 2.0 mg total), cyclophosphamide 750 mg/m^2 IV on Day 1 and oral or IV prednisone/prednisolone 100 mg on Day 1 to Day 5 of each 21 day treatment cycle for 6 to 8 cycles. Treatment continued until 6-8 cycles were completed, unless unacceptable toxicity, treatment change, disease progression, or withdrawal of consent, occurred first. An additional two doses (1 dose per 21-day cycle) of single agent rituximab after the 6 cycles of treatment were completed if considered standard of care per local practice.
Period: Pre-Treatment Period
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Started (Started = Randomized) | 285 | 285
Completed (Completed = Received StudyTreatment) | 284 | 283
Not Completed | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Participant withdrew consent | 1 | 0
Period: Treatment Period
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Started | 283 (1 participant was initially randomized in the Placebo plus R-CHOP Arm, but received lenalidomide, and thus, was reassigned to the R2-CHOP Arm.) | 284 (2 participants were initially randomized in the R2-CHOP Arm, they never received a dose of lenalidomide, and thus, were reassigned to the Placebo-R-CHOP Arm.)
Completed (Completed = six full cycles of both len/pbo and R-CHOP) | 211 | 240
Not Completed | 72 | 44

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population was defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP | Total
Number analyzed (Participants) | 285 | 285 | 570
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (11.72) | 63.9 (9.35) | 63.2 (10.62)
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 138 | 137 | 275
  ≥ 65 | 147 | 148 | 295
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 142 | 263
  Male | 164 | 143 | 307
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 31
  Not Hispanic or Latino | 270 | 267 | 537
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 173 | 183 | 356
  Asian | 101 | 89 | 190
  Black or African American | 2 | 3 | 5
  Other | 3 | 2 | 5
  Not Collected or Reported | 6 | 8 | 14
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Body surface area is the calculated surface of a human body. BSA is often considered a more accurate measure of metabolic mass than body weight, since it's less affected by irregular amounts of fat tissue.
  m^2 | 1.780 (0.2167) | 1.775 (0.2101) | 1.777 (0.2132)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: 0 = Fully active, no restrictions; 1 = Restricted activity but ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities; 3 = Limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, no self-care, confined to bed or chair; 5 = Dead
  Participants
    0 = Fully Active | 129 | 111 | 240
    1 = Restrictive but ambulatory | 104 | 118 | 222
    2 = Ambulatory but unable to work | 52 | 56 | 108
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min] — Creatinine is a waste product from the normal breakdown of muscle tissue. As creatinine is produced, it's filtered through the kidneys and excreted in urine. Doctors measure the blood creatinine level as a test of kidney function. Population: One creatinine clearance value is missing.
  mL/min
    number analyzed (Participants) | 285 | 284 | 569
    (all) | 92.08 (35.576) | 90.19 (31.040) | 91.14 (33.373)
International Prognostic Index (IPI) Score [Count of Participants; unit: Participants] — The IPI score is a clinical tool developed to aid in predicting the prognosis of patients with aggressive non-Hodgkin's lymphoma, including DLBCL. One point is assigned for each of the following risk factors: Age greater than 60 years, Stage III or IV disease, elevated serum lactate dehydrogenase (LDH), ECOG performance status of 2, 3, or 4, more than 1 extranodal site. The sum of the points allotted correlates with the following risk groups: Low risk (0-1 points) Low-intermediate risk (2 points) High-intermediate risk (3 points) High risk (4-5 points)
  Participants
    = 2 | 121 | 120 | 241
    ≥ 3 | 164 | 165 | 329
Presence of Bulky Disease [Count of Participants; unit: Participants]
  < 7.0 cm (Non-Bulky Disease) | 188 | 186 | 374
  ≥ 7.0 cm (Bulky Disease) | 97 | 99 | 196
Disease Stage of Diffuse Large B-Cell Lymphoma at Diagnosis [Count of Participants; unit: Participants] — The criteria for clinical stage (Ann Arbor staging) are as below: I: involvement of a single nodal region. II: involvement of 2 or more lymph node regions on the same side of the diaphragm. III: involvement of lymph node regions on both sides of the diaphragm. IV: disseminated involvement of 1 or more extra-lymphatic sites with or without associated lymph node involvement.
  Participants
    Stage I | 0 | 1 | 1
    Stage II | 37 | 32 | 69
    Stage III | 80 | 98 | 178
    Stage IV | 168 | 154 | 322

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS)
Description: Progression free survival was defined as the time (months) from the date of randomization to the date of disease progression or death (any cause), whichever occurred earlier and was assessed by the Independent Response Adjudication Committee (IRAC). Relapse from complete response (CR) was considered as disease progression throughout the study. Disease progression was determined based on the Revised Response Criteria for Malignant Lymphoma. The PFS analysis was based on the censoring rules using the Food and Drug Administration (FDA) Guidance. Participants who did not experience disease progression and who did not die before the clinical data cutoff date were censored at the date of last adequate response assessment.
Time Frame: From the date of randomization up to the data cut off date of 15 March 2019; median follow-up of 24.5 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
months | NA [NA to NA] — Median PFS and the upper and lower 95% confidence interval was not reached due to the low number of events. | NA [35.5 to NA] — Median PFS and the upper and lower 95% confidence interval was not reached due to the low number of events.
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.2864, Log Rank; Stratified by: IPI score (2 or ≥ 3), presence or absence of bulky disease (diameter of the lesion ≥ 7 cm or < 7 cm), and age (< 65 or ≥ 65 years); Hazard Ratio (HR) = 0.849, 95% CI 2-sided [0.632 to 1.140] — Hazard ratio was derived from Cox proportional hazard model adjusting for the 3 stratification factors

2. Secondary Outcome: Kaplan-Meier (K-M) Estimate of Event Free Survival (EFS)
Description: EFS was defined as the time (months) from randomization until occurrence of one of the following events, whichever occurred first: • Disease progression • Initiation of subsequent systemic anti-lymphoma therapy • Death due to any cause The assessment of EFS was conducted by the IRAC using the International Working Group (IWG) criteria for NHL. Pre-specified optional therapies such as the extra 2 doses of single agent rituximab after Cycle 6 or consolidation radiotherapy did not count as an EFS event (initiation of subsequent systemic anti-lymphoma therapy) if the decision to treat and the location to be treated was determined prior to randomization. Participants who did not experience any of the events defined in the categories above before the clinical data cutoff date were censored at date last known alive.
Time Frame: From the date of randomization up to the data cut off date of 15 March 2019; median follow-up was 24.5 months
Population: The ITT population was defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Months | NA [NA to NA] — Median EFS was not reached due to the low number of events. | NA [31.3 to NA] — Median EFS was not reached due to the low number of events.
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.7294, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.038, 95% CI 2-sided [0.802 to 1.344] — Hazard ratio was derived from Cox proportional hazard model adjusting for the 3 stratification factors

3. Secondary Outcome: K-M Estimate of Overall Survival (OS)
Description: Overall survival was assessed by the Independent Response Adjudication Committee (IRAC) and defined as time from randomization until death due to any cause. Participants who withdrew consent were censored at the time of withdrawal. Participants who were still alive before the clinical data cutoff date and participants who were lost to follow-up were censored at date last known alive.
Time Frame: From randomization until death due to any cause (up to approximately 86 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Months | NA [NA to NA] — Median OS and the upper and lower 95% confidence interval were not reached due to the low number of events. | NA [NA to NA] — Median OS and the upper and lower 95% confidence interval were not reached due to the low number of events.
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.8760, Log Rank; Log-rank test stratified by 3 factors: IPI score (2 or ≥ 3), presence of bulky disease (bulky or nonbulky), and age (< 65 or ≥ 65); Hazard Ratio (HR) = 0.965, 95% CI 2-sided [0.716 to 1.300] — Hazard ratio was derived from Cox proportional hazard model adjusting for the 3 stratification factors

4. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response (CR)
Description: The percentage of participants who achieved a CR after initiation of the study treatment and prior to initiation of subsequent systemic antilymphoma therapy as assessed by the IRAC. A CR = complete metabolic response; target nodes/nodal masses regressed on computed tomography to (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm prior to therapy. Regressed to normal size by imaging, and absence of nodules related to lymphoma. If bone marrow was involved prior to therapy, no evidence of fluorodeoxyglucose avid disease in marrow per International Working Group (IWG) 2014 for Non-Hodgkin's Lymphoma (NHL). Participants who did not have any adequate response assessments during this period were not considered as responders.
Time Frame: From randomization date up to the data cut off date of 15 March 2019; median follow-up was 24.5 months
Population: The ITT population was defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not. Participants who had a CR.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Percentage of Participants | 69.1 [63.4 to 74.4] | 64.9 [59.1 to 70.4]
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.2933, Cochran-Mantel-Haenszel — Obtained from CMH test adjusting for stratification factors: IPI score (2 or ≥ 3), presence of bulky disease (bulky or nonbulky), and age (< 65 or ≥ 65)

5. Secondary Outcome: Percentage of Participants Who Achieved an Objective Response
Description: An objective response = percentage of participants who achieved a complete response or partial response after initiation of the treatment and prior to initiation of subsequent systemic anti-lymphoma therapy. A CR = complete metabolic response; Target nodes/nodal masses regressed on computed tomography to (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm prior to therapy. Regressed to normal size by imaging, and absence of nodules related to lymphoma. If bone marrow was involved prior to therapy, no evidence of fluorodeoxyglucose avid disease in marrow. PR = ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. No increase in other nodes, liver, or spleen. Splenic nodules regressed by ≥ 50% in their SPD or for single nodules, in the greatest transverse diameter; no new lesions. Participants who did not have any adequate response assessments during this period were not considered as responders.
Time Frame: From randomization date up to the data cut off date of 15 March 2019; median total treatment duration was 18.10 weeks for both treatment arms; range = 1.6 to 29.0 weeks for R2-CHOP arm and 0.3 to 22.9 weeks for placebo-R-CHOP arm
Population: The Intent-to-treat population was defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not. Participants who had a PR or better.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Percentage of Participants | 90.9 [86.9 to 94.0] | 90.9 [86.9 to 94.0]
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.9964, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: K-M Estimate of Duration of Complete Response
Description: Duration of complete response was calculated for complete responders only and was defined as the time from documented initial complete response prior to initiation of subsequent systemic antilymphoma therapy until documented disease progression or death, whichever occurred earlier. Participants who had not progressed or died at the time of the analysis were censored at the date of last response assessment demonstrating no disease progression. Participants who changed treatment without evidence of disease progression were censored at the last assessment showing no progression prior to treatment change.
Time Frame: From randomization date up to the data cut off date of 15 March 2019; median follow-up was 24.5 months.
Population: The ITT population was defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not. Participants who had a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 197 | 185
Months | NA [NA to NA] — Median duration of CR could not be estimated due to the low number of events. | NA [NA to NA] — Median duration of CR could not be estimated due to due to the low number of events.
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.2143, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.521 to 1.157] — HR was derived from COX model adjusting for the 3 stratification factors mentioned above

7. Secondary Outcome: K-M Estimate of Time to Next Lymphoma Therapy (TTNLT)
Description: Time to next lymphoma therapy was defined as the time from randomization to the time of treatment change for the next lymphoma treatment. Participants without treatment change were censored at date last known alive. Pre-specified optional therapies such as the extra 2 doses of single agent rituximab after Cycle 6 or consolidation radiotherapy did not count as treatment change for the next lymphoma therapy if the decision to treat and the location to be treated were determined prior to randomization.
Time Frame: From randomization date up to the data cut off date of 15 March 2019; median follow-up was 24.5 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Months | NA [NA to NA] — Median time to next lymphoma treatment was not reached due to low number of events. | NA [NA to NA] — Median time to next lymphoma treatment was not reached due to low number of events.
Statistical Analysis 1: Comparison: Lenalidomide Plus R-CHOP (R2-CHOP) vs Placebo Plus R-CHOP; Test type: Superiority; p = 0.3150, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.167, 95% CI [0.856 to 1.590] — HR is derived from Cox model

8. Secondary Outcome: Percentage of Participants Who Completed the Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym) Questionnaire
Description: The completion rate for FACT-Lym assessments was judged by looking at the number of completed FACT-Lym assessments at each time point. The FACT-Lym was considered completed if at least 1 calculable score was present. Completion rates were calculated as the number and percentage of participants out of the total number of patients in the ITT population and summarized by visit/cycle and treatment group. The FACT-Lym is a health related quality of life (HRQoL) questionnaire targeted to the management of chronic illness, predominantly within oncology and is considered an extension of the FACT-General questionnaire.
Time Frame: Screening, Midcycle = after Cycle 3 but before Cycle 4, Cycle 6 Day 1 (C6D1), End of Treatment (C6,D21), and Follow-Up Period up to Week 34
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Percentage of Participants
  Screening | 98.6 | 98.2
  Midcycle = After Cycle 3, but before Cycle 4 | 87.0 | 86.3
  End of Treatment (EoT) = 3-4 weeks after C6 | 76.1 | 79.6
  Follow-Up Period: Week 34 | 67.7 | 69.5

9. Secondary Outcome: Percentage of Participants Who Completed the Euroqol 5-Dimension 3-Level (EQ-5D-3L) Health Related Quality of Life (HR-QoL) Questionnaire
Description: The completion rate for EQ-5D assessments was judged by looking at the number of completed assessments at each time point. Completion rates were calculated as the number and percentage of participants out of the total number of patients in the ITT population and summarized by visit/cycle and treatment group. The EQ-5D-3L is a generic, self-reported preference-based measure of health across five dimensions: mobility, self-care, pain, usual activities, and anxiety/depression. Each dimension has three levels of 'severity' corresponding to "no problems", "some problems" and "extreme problems". The instrument is scored using the United Kingdom (UK) index ranges from -0.594 - 1, where 0 equates to death and 1 equates to full health -0.594 is considered 'worse than death'.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 285 | 285
Percentage of Participants
  Screening | 98.9 | 97.9
  Midcycle | 87.0 | 86.3
  End of Treatment (EoT) | 76.5 | 79.6
  Follow-Up Period: Week 34 | 68.1 | 69.1

10. Secondary Outcome: Mean Change From Baseline in the FACT-Lym Physical Well-Being Subscale
Description: The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on HRQL and contains 42 questions covering HRQL and common lymphoma symptoms and treatment side-effects. It begins with the Functional Assessment of Cancer Therapy - General (FACT-G), which contains 27 questions covering four core subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 questions) used to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). The physical well-being subscale ranges from 0 to 28, where higher scores reflect better HRQoL.
Time Frame: Baseline and Midcycle = after Cycle 3 but before Cycle 4, Cycle 6 Day 1 (C6D1), End of Treatment (C6,D21), and Follow-Up Period up to Week 34
Population: The HRQoL evaluable population was defined as all participants in the ITT population who had: at least one baseline and the corresponding post-baseline calculable FACT-Lym score assessment; where post-baseline is any subsequent time excluding unscheduled visits (i.e. at Midcycle, C6D1, EOT or a follow-up visit).
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 257 | 257
Units on a Scale
  Midcycle: number analyzed (Participants) | 246 | 244
  Midcycle | -0.7 (5.91) | 0.2 (5.40)
  C6 D1: number analyzed (Participants) | 140 | 137
  C6 D1 | -0.0 (6.35) | 0.9 (6.02)
  EoT = 3-4 weeks after C6: number analyzed (Participants) | 214 | 226
  EoT = 3-4 weeks after C6 | 1.5 (5.53) | 0.7 (5.72)
  Follow-Up Period: Week 34: number analyzed (Participants) | 191 | 196
  Follow-Up Period: Week 34 | 2.8 (5.24) | 2.6 (5.55)

11. Secondary Outcome: Mean Change From Baseline in the FACT-Lym Additional Concerns Subscale
Description: The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on HRQL and contains 42 questions covering HRQL and common lymphoma symptoms and treatment side-effects. It begins with the Functional Assessment of Cancer Therapy - General (FACT-G), which contains 27 questions covering four core subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 questions) used to assess NHL-related symptoms such as pain, itching, night sweats,trouble sleeping, fatigue and trouble concentrating and concerns regarding lumps and swelling, fevers, infections, weight, appetite, emotional stability and treatment. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). The Additional Concerns subscale ranges from 0 to 60, where higher scores reflect better HRQoL.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 257 | 255
Units on a Scale
  Midcycle: number analyzed (Participants) | 244 | 242
  Midcycle | 3.8 (10.33) | 4.1 (8.88)
  C6 D1: number analyzed (Participants) | 139 | 135
  C6 D1 | 5.8 (11.11) | 5.2 (9.40)
  EoT = 3-4 weeks after C6: number analyzed (Participants) | 212 | 222
  EoT = 3-4 weeks after C6 | 6.6 (10.11) | 4.5 (9.62)
  Follow-Up Period: Week 34: number analyzed (Participants) | 189 | 195
  Follow-Up Period: Week 34 | 8.3 (10.61) | 6.5 (9.20)

12. Secondary Outcome: Mean Change From Baseline in the FACT-Lym Functional Well-Being Subscale
Description: The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on HRQL and contains 42 questions covering HRQL and common lymphoma symptoms and treatment side-effects. It begins with the Functional Assessment of Cancer Therapy - General (FACT-G), which contains 27 questions covering four core subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 questions) used to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). The functional well-being subscale ranges from 0 to 28, where higher scores reflect better HRQoL.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 258 | 256
Units on a Scale
  Midcycle: number analyzed (Participants) | 246 | 242
  Midcycle | -0.5 (6.12) | 0.5 (5.84)
  C6 D1: number analyzed (Participants) | 139 | 135
  C6 D1 | 0.0 (6.24) | 1.4 (5.63)
  EoT = 3-4 weeks after C6: number analyzed (Participants) | 214 | 224
  EoT = 3-4 weeks after C6 | 1.0 (6.53) | 0.7 (6.71)
  Follow-Up Period: Week 34: number analyzed (Participants) | 191 | 196
  Follow-Up Period: Week 34 | 2.3 (6.65) | 3.1 (6.17)

13. Secondary Outcome: Mean Change From Baseline in the FACT-Lym Trial Outcome Index (TOI)
Description: The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on HRQL and contains 42 questions covering HRQL and common lymphoma symptoms and treatment side-effects. It begins with the Functional Assessment of Cancer Therapy - General (FACT-G), which contains 27 questions covering four core subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 questions) used to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). The FACT-Lym TOI is calculated by summing the Physical Well-being, Functional Well-being and Additional Concerns scores and has a range of 0 to 116. Higher scores reflect better HRQoL or fewer symptoms.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 256 | 254
Units on a Scale
  Midcycle: number analyzed (Participants) | 244 | 240
  Midcycle | 2.6 (18.26) | 4.6 (16.49)
  C6 D1: number analyzed (Participants) | 138 | 133
  C6 D1 | 5.9 (19.85) | 7.5 (17.40)
  EoT = 3-4 weeks after C6: number analyzed (Participants) | 212 | 220
  EoT = 3-4 weeks after C6 | 9.1 (18.51) | 5.8 (18.64)
  Follow-Up Period: Week 34: number analyzed (Participants) | 189 | 193
  Follow-Up Period: Week 34 | 13.5 (18.74) | 12.2 (17.97)

14. Secondary Outcome: Mean Change From Baseline in the Euroqol 5-Dimension 3-Level (EQ-5D-3L) Index Score
Description: The EQ-5D-3L is a generic, self-reported preference-based measure of health across five dimensions: mobility, self-care, pain, usual activities, and anxiety/depression. Each dimension has three levels of 'severity' corresponding to "no problems", "some problems" and "extreme problems". The instrument is scored as a single summary index using one of the available EQ-5D-3L value sets; in this study the UK scoring weights 9 were used. The UK index ranges from -0.594 to 1, where 0 equates to death and 1 equates to full health (-0.594 is considered 'worse than death').
Time Frame: as for outcome 10
Population: The HRQoL evaluable population was defined as all participants in the ITT population who had: at least one baseline and the corresponding post-baseline calculable EQ-5D score assessment; where post-baseline is any subsequent time excluding unscheduled visits (i.e. at Midcycle, C6D1, EOT or a follow-up visit).
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 257 | 255
Units on a Scale
  Midcycle: number analyzed (Participants) | 245 | 241
  Midcycle | 0.08 (0.308) | 0.08 (0.281)
  C6 D1: number analyzed (Participants) | 139 | 135
  C6 D1 | 0.10 (0.325) | 0.14 (0.330)
  EoT = 3-4 weeks after C6: number analyzed (Participants) | 214 | 223
  EoT = 3-4 weeks after C6 | 0.10 (0.309) | 0.06 (0.319)
  Follow-Up Period: Week 34: number analyzed (Participants) | 190 | 195
  Follow-Up Period: Week 34 | 0.15 (0.293) | 0.09 (0.311)

15. Secondary Outcome: Mean Change From Baseline in the EQ-5D-3L Visual Analogue Scale (VAS)
Description: The EQ-5D-3L questionnaire includes a visual analogue scale which records the respondent's self-rated health on a vertical, 0-100 scale where 100 = "Best imaginable health state" and 0 = "Worst imaginable health state". Higher scores again indicate better HRQoL and positive change scores indicate that post screening values were higher than those observed at screening. The EQ-5D-3L is a generic, self-reported preference-based measure of health across five dimensions: mobility, self-care, pain, usual activities, and anxiety/depression. Each dimension has three levels of 'severity' corresponding to "no problems", "some problems" and "extreme problems".
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
Number analyzed (Participants) | 256 | 255
Units on a Scale
  Midcycle: number analyzed (Participants) | 245 | 242
  Midcycle | 4.0 (20.5) | 3.0 (18.2)
  C6 D1: number analyzed (Participants) | 138 | 135
  C6 D1 | 6.0 (23.5) | 9.0 (24.5)
  EoT = 3-4 weeks after C6: number analyzed (Participants) | 213 | 224
  EoT = 3-4 weeks after C6 | 8.0 (18.7) | 6.0 (21.5)
  Follow-Up Period: Week 34: number analyzed (Participants) | 190 | 195
  Follow-Up Period: Week 34 | 12.0 (20.2) | 9 (21.4)

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization until study completion (assessed up to approximately 86 months). SAEs and Other AEs were monitored from the participant's first dose of study treatment up to 28 days after their last dose of LEN/PBO or any component of R-CHOP including the optional 2 additional doses of rituximab; measured up to approximately 33 weeks.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants (ITT Population).
  Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication (Safety Population).
Arm/Group | Lenalidomide Plus R-CHOP (R2-CHOP) | Placebo Plus R-CHOP
All-Cause Mortality (participants affected / at risk) | 85/285 | 88/285
Serious Adverse Events (participants affected / at risk) | 104/283 | 88/284
Other Adverse Events (participants affected / at risk) | 272/283 | 270/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus R-CHOP (R2-CHOP) (N=283) | Placebo Plus R-CHOP (N=284)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 31 | 14
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 19 | 13
Splenic necrosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 4
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 2 | 1
Death (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 9
Sudden cardiac death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 2
Device related sepsis (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 15 | 9
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 2 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 4
Varicella (Infections and infestations) | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 2
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 2
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Tic (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus R-CHOP (R2-CHOP) (N=283) | Placebo Plus R-CHOP (N=284)
Anaemia (Blood and lymphatic system disorders) | 127 | 95
Leukopenia (Blood and lymphatic system disorders) | 50 | 50
Lymphopenia (Blood and lymphatic system disorders) | 35 | 31
Neutropenia (Blood and lymphatic system disorders) | 183 | 150
Thrombocytopenia (Blood and lymphatic system disorders) | 68 | 55
Abdominal pain (Gastrointestinal disorders) | 18 | 16
Abdominal pain upper (Gastrointestinal disorders) | 11 | 18
Constipation (Gastrointestinal disorders) | 92 | 81
Diarrhoea (Gastrointestinal disorders) | 49 | 40
Nausea (Gastrointestinal disorders) | 64 | 66
Stomatitis (Gastrointestinal disorders) | 33 | 37
Vomiting (Gastrointestinal disorders) | 32 | 26
Asthenia (General disorders) | 39 | 28
Fatigue (General disorders) | 40 | 50
Oedema peripheral (General disorders) | 33 | 32
Pyrexia (General disorders) | 52 | 40
Upper respiratory tract infection (Infections and infestations) | 23 | 18
Infusion related reaction (Injury, poisoning and procedural complications) | 27 | 30
Alanine aminotransferase increased (Investigations) | 32 | 27
Aspartate aminotransferase increased (Investigations) | 22 | 20
Lymphocyte count decreased (Investigations) | 16 | 12
Platelet count decreased (Investigations) | 21 | 10
Weight decreased (Investigations) | 21 | 10
White blood cell count decreased (Investigations) | 35 | 19
Decreased appetite (Metabolism and nutrition disorders) | 29 | 32
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 41 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 22
Dizziness (Nervous system disorders) | 16 | 16
Dysgeusia (Nervous system disorders) | 10 | 15
Headache (Nervous system disorders) | 26 | 28
Neuropathy peripheral (Nervous system disorders) | 19 | 12
Paraesthesia (Nervous system disorders) | 26 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 51 | 51
Insomnia (Psychiatric disorders) | 23 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 48 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02285062/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT02285062/SAP_001.pdf